CLINICAL TRIAL: NCT04293523
Title: A 48-Month, Multi-Centre, Observational Study to Evaluate Long-Term Effectiveness of Elocta on Joint Health
Brief Title: A 48-Month Study to Evaluate Long-Term Effectiveness of Elocta on Joint Health
Acronym: A-MORE
Status: Active, not recruiting | Type: Observational
Sponsor: Swedish Orphan Biovitrum (Industry)
Responsible Party: Sponsor
Other Study IDs: Sobi.Elocta-005
Record Dates: First submitted 2020-02-20; First posted 2020-03-03 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Hemophilia A
Keywords: Joint health; HEAD-US; HJHS
MeSH Terms: conditions — Hemophilia A | interventions — factor VIII-Fc fusion protein

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hemophilia A patients: All patients diagnosed with haemophilia A regardless of severity, on factor treatment with Elocta according to usual clinical practice.
  Interventions: Drug: ELOCTA

INTERVENTIONS:
Drug: ELOCTA — Extended half-life factor VIII product
  Other Names: ELOCTATE; efmoroctocog alfa; rFVIIIFc

SUMMARY:
This is a 48-month observational, prospective, multicentre study. The overall aim of the study is to evaluate the long-term effectiveness of Elocta treatment on joint health in patients treated prophylactically with Elocta in a real-world setting.

DETAILED DESCRIPTION:
Haemophilia A is a rare genetic disorder estimated to occur in one out of 10,000 live births, characterized by a deficiency in coagulation factor VIII causing impaired haemostasis and prolonged bleeding episodes. Moderate haemophilia, defined as < 5%, and severe haemophilia, defined as < 1% of normal factor VIII activity result in frequent and spontaneous bleeds into muscles and joints, commonly the elbows, knees, and ankles. Bleeding into joints can cause acute pain and swelling and can result in reduced joint range of motion, long-term cartilage damage and debilitating haemophilic arthropathy. Early use of prophylaxis with factor VIII replacement is recommended following diagnosis of haemophilia A to maintain joint health and prevent joint destruction. However, despite the use of prophylaxis many patients still experience joint bleeds which may lead to joint deterioration over time. The risk of joint bleeds increases with the amount of time spent below certain FVIII trough levels, e.g. 1, 3 or 5 IU/dL. Thus, there is probably a relation between the intensity of the prophylactic treatment regimen and joint health. Elocta is an extended half-life rFVIII product (EHL rFVIII), with a slower clearance as compared to conventional FVIII products. Treatment with Elocta will therefore provide the treater with a greater flexibility for individualizing prophylaxis as compared to conventional FVIII. Higher trough levels can be reached with Elocta without increasing factor usage or injection frequency. The treater can instead choose to reduce the injection frequency or the factor consumption without lowering trough levels.

Patients may limit their physical activities due to fear of bleeding if they are unaware of their current FVIII level. Patient apps and wearables are now available which allow patients to view their predicted FVIII levels, and capture health-related data (such as bleedings, pain, well-being, physical activity levels etc.). This data can be shared with the treating physician supporting the planning to individualize the patient's factor treatment based on current lifestyle, health status and physical activity levels. Florio, a certified medical device used as part of routine clinical practice, is such an app, and the data output and patient feedback on their activity levels and sense of protection while using Florio will be analysed as exploratory objectives in this study.

The main purpose of this study is to evaluate the effectiveness of Elocta on joint health over a long observation period (48 months). The study will also explore the influence on long term joint health of different Elocta prophylaxis regimens leading to different trough levels and if the extent of patients' physical activity levels can be associated with predicted FVIII levels.

ELIGIBILITY:
Inclusion Criteria:

* Provided signed and dated informed consent by the patient, or the patient's legally authorized representative(s) for patients under the legal age, before any study-related activities are undertaken. Assent should be obtained from paediatric patients according to local regulations
* Have a diagnosis of haemophilia A
* At enrolment on prophylactic treatment with Elocta, independent of participation in the study

Exclusion Criteria:

* Enrolment in another concurrent clinical interventional study, or intake of an Investigational Medicinal Product (IMP), within three months prior to inclusion in this study
* Presence of factor VIII antibodies (inhibitors) (≥0.60 Bethesda Unit [BU]/mL) at the latest available inhibitor test

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with haemophilia A regardless of severity, of any gender and age, on factor treatment with Elocta according to usual clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 427 (Actual)
Dates: Start 2020-03-30 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Joint health: Target joint development | 48 months
  Number of target joints
Joint health: Target joint resolution | 48 months
  Number of resolved target joints
Joint health: Target joint recurrence | 48 months
  Number of recurring target joints
Joint health: Annualised joint bleeding rate (AJBR) for treated bleeds | 48 months
  Number of joint bleeding events per year, for treated bleeds

SECONDARY OUTCOMES:
Disease Activity (hypertrophic synovium) and Disease Damage (Cartilage or Bone) scores for elbows, knees and ankles | 48 months
  The Haemophilia Early Arthropathy Detection with UltraSound (HEAD-US) protocol will be used. The total score represents the sum of item scores for abnormalities detected. Its values range from 0 (minimum) to 8 (maximum). A higher score indicates a worse outcome.
Global Gait Score, and/or joint score items for elbows, knees and ankles. | 48 months
  The Haemophilia Joint Health Score (HJHS) system will be used. Global Gait Score, and/or Joint score items (swelling, duration of swelling, muscle atrophy, axial alignment, crepitus on motion, flexion loss, instability, extension loss, joint pain, strength, gait) for elbows, knees and ankles.
  The minimum score per joint is 0, the maximum score is 20. The overall total joint score (range 0-120) is the sum of the 6 six index joint (elbows, knees and ankles) scores. A higher score indicates a worse outcome.
Joint and physical evaluation for elbows, knees and ankles. | 48 months
  The WFH Physical Examination Score (AKA Gilbert Score) will be used. Joint evaluation (pain, bleeding, physical examination and radiologic evaluation) and physical evaluation (swelling, muscle atrophy, axial deformity, crepitus on motion, range of motion, flexion contracture, and instability). A higher score indicates a worse outcome.

OTHER OUTCOMES:
Effectiveness of Elocta: Annualised bleeding rate (ABR) for treated bleeds | 48 months
  Number of bleeding events per year, for treated bleeds
Effectiveness of Elocta: Annualised bleeding rate (ABR) for all bleeds | 48 months
  Number of bleeding events per year, for all bleeds
Effectiveness of Elocta: Occurrence of zero (0) joint bleeds | 48 months
  Percentage (%) of study population with zero (0) joint bleeds
Effectiveness of Elocta: Work productivity and impairment | 48 months
  Assessed by WPAI-SHP questionnaire
Effectiveness of Elocta: Quality of Life | 48 months
  Assessed by Haemo-QoL/Haem-A-QoL questionnaire
Effectiveness of Elocta: Physical activity level | 48 months
  Assessed by the Saltin-Grimby scale
Effectiveness of Elocta: Quality of Life | 48 months
  Assessed by EQ-5D-5L/EQ-5D-Y questionnaire
Effectiveness of Elocta: Severity of joint health | 48 months
  Assessed by Patient Global Impression of Severity of Joint Health questionnaire
Effectiveness of Elocta: FVIII plasma levels | 48 months
  Percentage (%) of FVIII plasma level
Effectiveness of Elocta: Usage of pain and anti-inflammatory medication | 48 months
  Assessed by medication dose
Effectiveness of Elocta: Usage of pain and anti-inflammatory medication | 48 months
  Assessed by total number of exposure days per medication
Usage of Elocta: Annualised injection frequency per subject | 48 months
  Assessed by prescription
Usage of Elocta: Annualised factor consumption per subject | 48 months
  Assessed by prescription [IU/kg]
Usage of Elocta: Adherence | 48 months
  Investigator assessed (Percentage (%))
Exploratory Objective | 48 months
  Influence of different Elocta prophylaxis regimens on long term joint health
Exploratory Objective: Impact of florio HAEMO on patients' sense of protection and their activity level | 48 months
  Results from questionnaire on impact of florio HAEMO tools on patients' sense of protection and their activity level
Exploratory Objective: Explore adherence to prescribed treatment regimen | 48 months
  florio HAEMO captured treatment adherence scores
Exploratory Objective: Explore relationship between predicted FVIII levels and physical activity | 48 months
  florio HAEMO captured predicted FVIII levels, florio HAEMO captured physical activity (type, duration, heart rate and steps)
Exploratory Objective: Explore timing of bleeds in relation to predicted FVIII levels and physical activity | 48 months
  florio HAEMO captured bleed data (timing, location, cause, treated/untreated), florio HAEMO captured injection data (time, dose), florio HAEMO captured predicted FVIII levels
Exploratory Objective: Explore the use of Florio to characterise pain and well-being | 48 months
  florio HAEMO captured pain data (time, location, cause, intensity), florio HAEMO captured well-being data
Exploratory Objective: Influence of different Elocta prophylaxis regimens on long term joint health | 48 months
  Target joint development, resolution and recurrence
Exploratory Objective: Influence of different Elocta prophylaxis regimens on long term joint health | 48 months
  Annualised joint bleeding rate (AJBR) for treated bleeds
Exploratory Objective: Influence of different Elocta prophylaxis regimens on long term joint health | 48 months
  Ultrasound (HEAD-US)
Exploratory Objective: Influence of different Elocta prophylaxis regimens on long term joint health | 48 months
  Clinical joint scoring (HJHS)
Exploratory Objective: Influence of different Elocta prophylaxis regimens on long term joint health | 48 months
  Annualised bleeding rate (ABR) (based on bleeding episodes assessed according to local practice) for all bleeds
Exploratory Objective: Influence of different Elocta prophylaxis regimens on long term joint health | 48 months
  Occurrence of zero (0) joint bleeds
Exploratory Objective: Influence of different Elocta prophylaxis regimens on long term joint health | 48 months
  Quality of Life assessed by Haemo-QoL/Haem-A-QoL
Exploratory Objective: Influence of different Elocta prophylaxis regimens on long term joint health | 48 months
  Physical activity level assessed by the Saltin-Grimby scale

CONTACTS AND LOCATIONS:
Overall Officials: Study Physician, Study Director — Swedish Orphan Biovitrum AB
Locations (53):
- Czechia (3):
  - University Hospital Brno, Brno
  - University Hospital Ostrava, Ostrava
  - Dept. of Pediatric Haematology and Oncology, University Hospital Motol, Prague
- Estonia (2):
  - Lastehaigla, Tallinn (Tallinn Children´s Hospital), Tallinn
  - The North Estonia Medical Centre Hematoloogiakeskus, Regionalhaigla, Tallinn
- Finland (2):
  - Helsinki University Central Hospital, New Children Hospital, Helsinki
  - Turku University Central Hospital, Paediatric and adolescent haematology and oncology clinic, Turku
- Germany (10):
  - Charité-Universitätsmedizin Berlin Campus Virchow Klinikum, Berlin
  - Universitätsklinikum Bonn AöR, Institut für Experimentelle Hämatologie und Transfusionsmedizin, Bonn
  - Hämostaseologie/Hämophiliezentrum, Medizinische Klinik 2 Institut für Transfusionsmedizin, Universitätsklinikum, Frankfurt
  - Universitätsklinikum Frankfurt - Klinik für Kinder- und Jugendmedizin, Frankfurt
  - Universitätsklinikum Hamburg-Eppendorf (UKE), Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Werlhof-Institut für Hämostaseologie GmbH, Hanover
  - SRH-Klinikum Heidelberg, Heidelberg
  - HZRM Hämöphilie Zentrum Rhein Main, Mörfelden-Walldorf
  - Kinderklinik und Kinderpoliklinik im Dr. von Haunerschen Kinderspital am Universitätsklinikum München, München
- Greece (2):
  - Ippokrateio Hospital Thessaloniki (adult department), Thessaloniki
  - Ippokrateio Hospital Thessaloniki (pediatric department), Thessaloniki
- Italy (7):
  - University of Bari Aldo Moro (Centro Emofilia Policlinico - Pediatria U.O.), Bari
  - AUSL Romagna Centro Emofilia U.O.C., Medicina Trasfusionale Dipartimento Patologia, Clinica Ospedale M. Bufalini, Cesena
  - Giannina Gaslini Institute, Genova
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan
  - University Hospital of Parma, AOUP, Haemophilia Center, Parma
  - Uo Malattie Emorragiche e Trombotiche Fondazione Policlinico Universitario Agostino Gemelli, IRCCS, Universitá Catolica del Sacro Coure, Rome
  - Azienda Ospedaliera Città della Salute e della Scienza di Torino Regina Margherita, Torino
- University Medical Center Groningen/UMCG, Groningen, Netherlands
- The Royal Hospital, Muscat, Oman
- Saudi Arabia (4):
  - Dr Suliman Al Habib Hospital Riyadh, Riyadh
  - King Faisal Specialised Hospital, KFSH Riyadh, Children, Riyadh
  - King Faisal Specialist Hospital KFSH, Adults, Riyadh
  - Riyadh Military Hospital (P.S.M.C), Riyadh
- University Medical Centre Ljubljana Division of Paediatrics, Ljubljana, Slovenia
- Spain (12):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Sant Johan De Deu, Barcelona
  - Hospital Universitario Cruces, Cruces
  - Hospital Universitario Donostia, Donostia / San Sebastian
  - Hospital Universitario Carlos Haya, Málaga
  - Hospital Virgen de la Arrixaca, Murcia
  - Complejo Hospitalario de Navarra, Navarro
  - Hospital Universitario Central de Asturias (HUCA), Oviedo
  - Hospital Universitario Son Espases, Palma de Mallorca
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Alvaro Cunqueiro, Vigo
- Sweden (2):
  - Hematologimottagning Sahlgrenska, Gothenburg
  - Department of Haematology, Oncology and Radiation Physics, Skåne University Hospital Malmö, Malmo
- Switzerland (4):
  - Universitätsklinik für Hämatologie und Hämatologisches Zentrallabor Inselspital, Bern
  - Service et Laboratoire central d'hématologie, Adults, Lausanne
  - Zentrum für Labormedizin, Sankt Gallen
  - Universitätsspital Zürich Klinik für Medizinische Onkologie und Hämatologie, Zurich
- United Kingdom (2):
  - East Kent Hospitals University NHS Foundation Trust, Kent Haemophilia and Thrombosis Centre, Kent and Canterbury Hospital, Canterbury
  - Great Ormond Street Hospital, Royal London Hospital for Integrated Medicine, London

IPD SHARING:
Plan to Share IPD: No